CLINICAL TRIAL: NCT04806035
Title: A Phase 1b Multi-cohort Study of TG-1801 Alone or in Combination With Ublituximab in Subjects With B-Cell Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: Study of TG-1801 Alone or in Combination With Ublituximab in Subjects With B-Cell Lymphoma or Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic/Business Decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-1801-102
Record Dates: First submitted 2021-03-05; First posted 2021-03-19 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: CLL; SLL; Richter's Transformation; Indolent Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Aggressive Lymphoma; DLBCL; Mediastinal Large B-cell Lymphoma; MCL
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — ublituximab; LFB-R603

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: TG-1801 (Experimental): TG-1801 Single Agent
  As per protocol v3.0, Cohort A is no longer enrolling.
  Interventions: Biological: TG-1801
- Cohort B: TG-1801 (Experimental): TG-1801 Single Agent, escalating doses
  Interventions: Biological: TG-1801
- Cohort C: TG-1801 + Ublituximab (Experimental): TG-1801 in combination with ublituximab
  As per protocol v3.0, ublituximab will be discontinued and the Cohort C is no longer enrolling.
  Interventions: Biological: TG-1801; Biological: Ublituximab

INTERVENTIONS:
Biological: TG-1801 — It is a bispecific, first-in-class, CD47 and CD19 antibody
  Other Names: NI-1701
Biological: Ublituximab — recombinant chimeric anti-CD20 monoclonal antibody, available in 25 mg/mL administered as an IV infusion once every 4 weeks
  Other Names: TG-1101; LFB-R603
  Arms: Cohort C: TG-1801 + Ublituximab

SUMMARY:
The primary objective of this study is to determine the recommended phase 2 dose (RP2D) and characterize the safety profile of TG-1801. As per protocol v3.0, ublituximab will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* B-cell non-Hodgkin lymphoma (NHL) including Richter's Transformation (RT) and transformed follicular lymphoma (FL), that warrants systemic therapy
* Chronic Lymphocytic Leukemia (CLL), that warrants systemic therapy as defined by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) (Hallek 2018)
* Treatment Status:

  1. NHL subjects: relapsed to or refractory after at least two prior standard systemic therapies (excluding antibiotics)
  2. RT subjects: relapsed or refractory after at least two prior lines of therapy for CLL/ Small lymphocytic lymphoma (SLL) or RT
  3. CLL subjects: relapsed to or refractory after at least two prior standard therapies
* Measurable disease defined as:

  1. NHL (including SLL): at least 1 measurable disease lesion > 1.5 centimeters (cm)
  2. CLL: at least 1 measurable disease lesion

Exclusion Criteria:

* Prior therapy with any agent blocking the CD47/SIRPα pathway or any previous CD19 targeting therapy,
* Subjects receiving cancer therapy (i.e. chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization) or any investigational drug within 21 days of Cycle 1 Day 1.
* Prior autologous stem cell transplant (SCT) within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
RP2D | Up to 24 months
  To determine the recommended Phase 2 dose (RP2D)

SECONDARY OUTCOMES:
Overall Response Rate | Up to 24 months
  To evaluate the overall response rate (ORR) of TG-1801

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - TG Therapeutics Investigational Trial Site, Fayetteville, Arkansas
  - TG Therapeutics Investigational Trial Site, Hackensack, New Jersey
  - TG Therapeutics Investigational Trial Site, Chattanooga, Tennessee
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Houston, Texas

REFERENCES:
- [Derived] Chauchet X, Cons L, Chatel L, Daubeuf B, Didelot G, Moine V, Chollet D, Malinge P, Pontini G, Masternak K, Ferlin W, Buatois V, Shang L. CD47xCD19 bispecific antibody triggers recruitment and activation of innate immune effector cells in a B-cell lymphoma xenograft model. Exp Hematol Oncol. 2022 May 10;11(1):26. doi: 10.1186/s40164-022-00279-w. PMID 35538512